CLINICAL TRIAL: NCT04195568
Title: EndoVascular Treatment Of Wide-Neck Aneurysms, an EvaLuation of Safety and EffectiVeness of Stryker Surpass Evolve™ Flow Diverter System
Brief Title: Evaluation of Safety and Effectiveness of Stryker Surpass Evolve™ Flow Diverter System
Acronym: EVOLVE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stryker Neurovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDM10001444
Record Dates: First submitted 2019-12-04; First posted 2019-12-12 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2024-11

CONDITIONS: Aneurysm, Intracranial
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Surpass Evolve Flow Diverter System (Experimental): This is a prospective single arm study in which all subjects who present for flow diverter implantation, provide informed consent, and meet inclusion/exclusion criteria may receive treatment (Surpass Evolve Flow Diverter).
  Interventions: Device: Surpass Evolve Flow Diverter System

INTERVENTIONS:
Device: Surpass Evolve Flow Diverter System — The Surpass Evolve Flow Diverter System is indicated for the endovascular treatment of adults (age 18 or above) with unruptured saccular wide-neck or fusiform intracranial aneurysms ≤12 mm.

SUMMARY:
The primary objective of this study is to evaluate the safety and effectiveness of the Surpass™ Evolve Flow Diverter System in the treatment of unruptured, wide-neck intracranial aneurysms measuring ≤ 12 mm and located on the ICA or its branches

DETAILED DESCRIPTION:
The Surpass Evolve Flow Diverter System is indicated for the endovascular treatment of adults (age 18 or above) with unruptured saccular wide-neck or fusiform intracranial aneurysms ≤ 12 mm for treatment in vessel diameters between 1.75-5.0mm.

ELIGIBILITY:
Inclusion Criteria:

1. Age is ≥ 18 and ≤ 80 years
2. Has a single unruptured target intracranial aneurysm (IA) with the following characteristics:

   1. Is located on the internal carotid artery (ICA) or its branches.
   2. Has a neck ≥ 4 mm, dome to neck ratio ≤ 2.0, or no discernible neck
   3. Aneurysm size is ≤ 12 mm (saccular or fusiform configuration)
3. Has a parent vessel diameter ≥ 1.75 mm and ≤ 5.0 mm at both the proximal and distal segments where the implant will be placed
4. Has multiple increased risk factors for intracranial (IA) aneurysm rupture, including but not limited to, aneurysm morphology, smoking, hypertension, diabetes, age, prior and/or family history of rupture, and/or history of subarachnoid hemorrhage that may result in a benefit risk profile of endovascular treatment that outweighs the risks of intracranial aneurysm rupture during the subject's expected lifetime if left untreated.

Exclusion Criteria:

1. Has an extradural target aneurysm
2. Has a target aneurysm in the posterior circulation
3. Perforator or branch vessel, inclusive of the posterior communicating artery, arises from the target aneurysm body or neck (branches or arteries must arise or connect from the parent vessel separate from the aneurysm or neck to not be excluded from study)
4. Has a true bifurcation aneurysm, defined as an aneurysm (saccular or non-saccular) located at a point of vessel bifurcation
5. Target aneurysm is unsuitable for flow diverter treatment
6. Has vessel characteristics, such as severe tortuosity (cICA Type IV), stenosis (>70%), or morphology that would preclude safe endovascular access to the target aneurysm necessary for treatment with the study device
7. Received previous treatment of the target aneurysm or parent artery where it would interfere with the placement or proper apposition of the device
8. Has a medical contraindication to study or procedure related antiplatelet medications (aspirin, clopidogrel/Plavix, ticagrelor, and heparin), local or general anesthesia, or life-threatening allergy to contrast dye
9. Has a known severe allergy to nickel, chromium cobalt, tungsten or platinum.
10. Modified Rankin Score (mRS) assessment is ≥ 3 at preprocedure exam
11. Presence of unstable neurological deficit (i.e., worsening of clinical condition in the last 30 days)
12. Subarachnoid hemorrhage occurred within 30 days prior to enrollment
13. Major surgery (including previous intracranial implant) occurred within previous 30 days or is planned in the next 120 days after enrollment date
14. Has more than one IA that requires treatment within 12 months
15. Received previous intracranial implant associated with the symptomatic or vascular distribution within the past 12 weeks prior to treatment date
16. Chronic anticoagulation therapy is ongoing or known coagulopathy exists
17. Has other known serious concurrent medical conditions such as heart disease (e.g., unstable atrial fibrillation [with or without pacemaker], recent myocardial infarction [< 12 weeks ago], symptomatic congestive heart failure, or carotid stenosis), kidney failure [>2.0mg/dl serum creatinine], pulmonary disease, uncontrolled diabetes, progressive neurologic disorders, terminal cancer, vasculitis, high risk of ischemic stroke or recent stroke
18. Has acute life-threatening illness other than the neurological disease (e.g., acute kidney or heart failure) to be treated in this trial
19. Life expectancy is less than 5 years due to other illness or condition (in addition to an intracranial aneurysm)
20. Unable to complete study follow up due to dementia or psychiatric problem, substance abuse, or history of noncompliance with medical advice
21. Pregnancy at time of enrollment
22. Presence of intracranial mass (tumor, except meningioma, abscess, or other infection), non-treated arteriovenous malformation (AVM) in the territory of the target aneurysm
23. Evidence of active infection at the time of treatment
24. Enrollment in another trial involving an investigational product that could confound the outcomes of this trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2024-09-11 (Actual); Study Completion 2028-09-13 (Estimated)

PRIMARY OUTCOMES:
Primary Effectiveness Endpoint | 12 months (± 3 months) post procedure
  The primary effectiveness endpoint of this study is a composite of 100% occlusion (Raymond 1, complete occlusion) of the target aneurysm without significant parent artery stenosis (>50% stenosis), per independent core lab assessment of digital subtraction angiography (DSA) images acquired at 12 months (± 3 months) post-procedure, and with no target aneurysm retreatment.
Primary Safety Endpoint | 12 Months (± 3 months) post procedure
  The primary safety endpoint of this study is neurologic death, or disabling stroke at 12 months as adjudicated by an independent Clinical Events Committee (CEC).

SECONDARY OUTCOMES:
Secondary Safety Endpoints | 3 Year Follow-Up
  The secondary safety endpoints will be evaluated throughout the study, and are as follows:
  1. Neurological death or major ipsilateral stroke as adjudicated by an independent Clinical Events Committee.
  2. Stroke in the treated vascular territory as adjudicated by a Clinical Events Committee

CONTACTS AND LOCATIONS:
Overall Officials: Adam S Arthur, MD, Principal Investigator — Semmes Murphy Clinic; Vitor M Pereira, MD, Principal Investigator — University Health Network, Toronto
Locations (37):
- United States (32):
  - DIGNITY HEALTH/ Barrow Neurological Institute, Phoenix, Arizona
  - St. Joseph's Hospital, Tucson, Arizona
  - University of California, Los Angeles, Los Angeles, California
  - Lyerly Baptist, Inc./Baptist Medical Center - Jacksonville/Lyerly Neurosurgery, Jacksonville, Florida
  - Mayo Clinic Florida, Jacksonville, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - Tallahassee Neurological Clinic, Tallahassee, Florida
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Baptist Healthcare System, Inc./Baptist Health, Lexington, Kentucky
  - Maine Medical Center, Portland, Maine
  - Tufts Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Lahey Clinic, Burlington, Massachusetts
  - University of Massachusetts, North Worcester, Massachusetts
  - Spectrum Health, Grand Rapids, Michigan
  - Robert Wood Johnson University Medical Center, New Brunswick, New Jersey
  - University of Buffalo, Buffalo, New York
  - ICAHN School of Medicine at Mount Sinai, New York, New York
  - Stony Brook, Stony Brook, New York
  - Montefiore Medical Center, The Bronx, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Geisinger Clinic, Wilkes-Barre, Pennsylvania
  - Semmes Murphey Clinic/ University of Tennessee Health Sciences Center, Memphis, Tennessee
  - University of Texas Medical Branch, Galveston, Texas
  - Valley Baptist Health System, Harlingen, Harlingen, Texas
  - University of Utah, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia
- Australia (3):
  - Liverpool Hospital, Liverpool, New South Wales
  - Sir Charles Gairdner Hospital, Nedlands, Perth
  - Gold Coast Hospital & Health Service/ Gold Coast University Hospital, Southport, Queensland
- Canada (2):
  - St. Michael's Hospital - Toronto, Toronto, Ontario
  - University Health Network/ Toronto Western Hospital, Toronto, Ontario